CLINICAL TRIAL: NCT03127605
Title: Inotuzumab Ozogamicin - PF-05208773
Status: Approved for marketing | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B193
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

MeSH Terms: interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin
  Other Names: PF-05208773

SUMMARY:
Inotuzumab Ozogamicin Expanded Access Program

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult